CLINICAL TRIAL: NCT00374634
Title: Individual Versus Standard rFSH Dose for Controlled Ovarian Stimulation and Intrauterine Insemination. A Prospective Randomised Multi Centre Study
Brief Title: Individual Versus Standard Follicle Stimulating Hormone Dose for Controlled Ovarian Stimulation and Insemination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nina la Cour Freiesleben (Other)
Responsible Party: Sponsor-Investigator, Nina la Cour Freiesleben, MD PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: indvFSH2006
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Individual" or "standard" rFSH dose (Active Comparator): Patients were randomized to recieve "individual" (50, 75 or 100 IU/day) or "standard" (75 IU/day) rFSh dose. The individual dose was prescribed according to a dosage nomogram based on the patient's body weight (kg) and the total antral follicle count (Freiesleben NC et al., RBMOnline 2009;17:632-64).
  Interventions: Drug: rFSH drug dose
- "Standard" rFSH dose (Active Comparator): "Standard" dose of rFSH
  Interventions: Drug: "Standard" rFSH dose

INTERVENTIONS:
Drug: rFSH drug dose — "Individual" rFSH dose (50, 75 or 100 IU rFSH/day)
  Arms: "Individual" or "standard" rFSH dose
Drug: "Standard" rFSH dose — "Standard" rFSH dose was 75 IU/day
  Arms: "Standard" rFSH dose

SUMMARY:
The purpose of this study is to test if recombinant follicle stimulating hormone (rFSH) given in individual doses, according to a nomogram we have constructed based on our results from a previous study, results in more patients maturing 2-3 follicles compared to standard dose.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-39 years
* First stimulation with rFSH only
* Indication for intrauterine insemination with standard rFSH starting dose
* Regular menstrual bleeding with a cycle between 21-35 days
* Two ovaries
* Bilateral tuba patency
* Semen analysis must be sufficient for insemination according to the diagnostic analysis.

Exclusion Criteria:

* More than three former stimulated intrauterine insemination cycles

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number of mature follicles in the study and control group.

SECONDARY OUTCOMES:
Number of cycles where the rFSH dose is changed.
Number of cycles cancelled or converted to in vitro fertilisation.
Pregnancy rate. | October 2008

CONTACTS AND LOCATIONS:
Overall Officials: Anders N Andersen, Professor,MD, Study Director — The Fertility Clinic, dep.4071, Copenhagen University Hospital, Rigshospitalet, Blegdamsvej 9, 2100 Copenhagen East, Denmark
Locations (1):
- The Fertility Clinic, dep.4071, Copenhagen University Hospital, Rigshospitalet, Copenhagen East, Denmark

REFERENCES:
- [Background] la Cour Freiesleben N, Lossl K, Bogstad J, Bredkjaer HE, Toft B, Rosendahl M, Loft A, Bangsboll S, Pinborg A, Nyboe Andersen A. Individual versus standard dose of rFSH in a mild stimulation protocol for intrauterine insemination: a randomized study. Hum Reprod. 2009 Oct;24(10):2523-30. doi: 10.1093/humrep/dep239. Epub 2009 Jul 14. PMID 19602518
- [Derived] Freiesleben Nl, Rosendahl M, Johannsen TH, Lossl K, Loft A, Bangsboll S, Friis-Hansen L, Pinborg A, Andersen AN. Prospective investigation of serum anti-Mullerian hormone concentration in ovulatory intrauterine insemination patients: a preliminary study. Reprod Biomed Online. 2010 May;20(5):582-7. doi: 10.1016/j.rbmo.2010.02.007. Epub 2010 Feb 12. PMID 20303323